CLINICAL TRIAL: NCT03877042
Title: The Efficacy of Using CR and PS Prosthesis in Total Knee Replacement: a Randomized, Double-blind, Controlled Trial
Brief Title: The Efficacy of Using CR and PS Prosthesis in Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Yanzhao, Principal Investigator, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJ2018004
Record Dates: First submitted 2019-03-06; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; CR; PS
MeSH Terms: interventions — Prostheses and Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental (Experimental): Patients with end-stage knee disease need Total Knee Arthroplasty in both knees.
  Interventions: Device: Cruciate-retaining (CR) prostheses; Device: Posterior-stabilized (PS) prostheses

INTERVENTIONS:
Device: Cruciate-retaining (CR) prostheses — One leg is conducted TKA with Cruciate-retaining (CR) prostheses.
Device: Posterior-stabilized (PS) prostheses — One leg is conducted TKA with Posterior-stabilized (PS) prostheses.

SUMMARY:
The investigators will investigate the efficacy of using CR and PS implants in TKA. The investigators will conduct TKA with different implants simultaneously on one patient to compare the post-operation efficacy of both implants.

DETAILED DESCRIPTION:
A randomized, single-center, single group study comparing the efficacy and safety of using CR and PS implants in TKA. The investigators will conduct TKA with different implants simultaneously on one patient to compare the post-operation efficacy of both implants. Subjects will be monitored through postoperative follow-up to understand the bilateral knee condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who plan to undergo primary total knee arthroplasty on bilateral knee joint with a diagnosis of osteoarthritis or rheumatoid arthritis, etc.;

Exclusion Criteria:

* Those who do not meet the inclusion criteria;
* Neuromuscular dysfunction;
* Diseases affecting postoperative efficacy evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
HSS score changes after TKA | 1,3,6,12 months after TKA
  Summed Hospital for special surgery (HSS) score with a maximum score of 100. Higher values represent a better outcome.
KSS score changes after TKA | 1,3,6,12 months after TKA
  Summed Knee Society Score (KSS) score with a maximum score of 100. Higher values represent a better outcome.
X-ray evaluation changes after TKA | 1,3,6,12 months after TKA
  Evaluation of postoperative X-ray results for lower limb line, prosthesis location and other conditions
Muscle strength measurement changes after TKA | 1,3,6,12 months after TKA
  Strength measurement of related muscles according to Lovett muscle strength grading standard.

CONTACTS AND LOCATIONS:
Overall Officials: Qingsheng Zhu, MD, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, China